CLINICAL TRIAL: NCT07213635
Title: Effect of Paracervical Block on Postoperative Opioid Use in Vaginal Hysterectomy for Prolapse: a Randomized, Placebo-Controlled Trial
Brief Title: Paracervical Injection and Opioid Use After Vaginal Hysterectomy for Prolapse
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 25-0619
Record Dates: First submitted 2025-10-02; First posted 2025-10-09 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Opioid Use; Surgical Recovery; Vaginal Hysterectomy; Prolapse Pelvic; Postoperative Pain
Keywords: paracervical block; vaginal hysterectomy; prolapse repair; postoperative opioid use; postoperative pain scores; postoperative recovery
MeSH Terms: conditions — Pain, Postoperative | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Paracervical block (Experimental): Participants randomized to this experimental arm will receive a paracervical block with 0.5% bupivacaine with epinephrine at the time of vaginal hysterectomy with prolapse repair
  Interventions: Drug: Bupivacaine-epinephrine
- Placebo (Placebo Comparator): Participants randomized to this experimental arm will receive a placebo paracervical injection with normal saline at the time of vaginal hysterectomy with prolapse repair
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Bupivacaine-epinephrine — Participants randomized to this experimental arm will receive a paracervical block with 10 mL 0.5% bupivacaine with epinephrine before their vaginal hysterectomy and prolapse repair
  Arms: Paracervical block
Drug: Normal saline — Participants randomized to this experimental arm will receive a placebo paracervical injection with 10 mL 0.5% normal saline before their vaginal hysterectomy and prolapse repair
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The goal of the study to see if giving a numbing medicine around the cervix (called a paracervical block) during vaginal hysterectomy with prolapse repair helps people feel less pain and need fewer strong pain medicines afterward.

The main question it aims to answer is:

• Does receiving a paracervical block at the time of vaginal hysterectomy with prolapse repair reduce postoperative opioid use?

Researchers will compare opioid use in participants who receive the an injected numbing medicine (bupivacaine with lidocaine) to those that receive a saltwater liquid placebo.

Participants will:

* Receive either an injection of the numbing medicine (bupivacaine with lidocaine) or saltwater liquid placebo after they are asleep but before any other parts of the surgery are done
* Record and report pain medications used for 7 days after surgery
* Report pain scores before discharge from the post anesthesia recovery area on day of surgery as well as 1 and 7 days after surgery
* Complete a surgical recovery questionnaire during 6 week postoperative visit
* Complete a one page multiple-choice test on pelvic organ prolapse

DETAILED DESCRIPTION:
Secondary outcomes are to:

1. Compare postoperative pain scores in patients undergoing vaginal hysterectomy for prolapse repair who receive an intraoperative paracervical block compared to placebo
2. Compare surgical recovery times in patients undergoing vaginal hysterectomy for prolapse repair who receive an intraoperative paracervical block compared to placebo.
3. Examine incidence of adverse events in patients undergoing vaginal hysterectomy for prolapse repair who receive intraoperative paracervical block compared to placebo

ELIGIBILITY:
Inclusion Criteria:

* Individuals undergoing vaginal hysterectomy with concomitant prolapse repair procedure

Exclusion Criteria:

* Non-English speaking
* Weight less than 50 kg
* Allergy to bupivacaine
* Pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-10-20 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative opioid use | Assessed verbally during a 5 minute phone call on day 1 and 7 following surgery
  Mean postoperative opioid use converted to morphine milligram equivalents

SECONDARY OUTCOMES:
Pain score | Assessed verbally prior to discharge from post anesthesia recovery area, and during 5 minute phone call on day 1 and 7 following surgery
  Mean numeric visual analog pain score from 0-10 where 0 is "no pain" and 10 is "worst pain you can imagine"
Global Surgical Recovery score | Assessed verbally during 5 minute phone call on day 1 and 7 following surgery.
  Mean Global Surgical Recovery score (from 0-100%) where 0% is not recovered at all and 100% is fully recovered.
Postdischarge Surgical Recovery | Assessed during completion of 5 minute survey on week 6 postoperative visit.
  Mean Postdischarge Surgical Recovery score (from 0-100) where higher scores denote better recovery.
Adverse events | From day of surgery until week 6 postoperative visit
  Number of hospital admission (including on day of surgery) and emergency department presentations as well as additional calls or urgent clinic visits

CONTACTS AND LOCATIONS:
Overall Officials: Bertie Geng, MD, Principal Investigator — University of North Carolina
Locations (1):
- University of North Carolina Urogynecology and Reconstructive Pelvic Surgery at REX, Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 12 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Time Frame: beginning 12 months following publication until 36 months following publication
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.